CLINICAL TRIAL: NCT03395587
Title: Phase II Trial of Vaccination with Lysate-loaded, Mature Dendritic Cells Integrated Into Standard Radiochemotherapy in Newly Diagnosed Glioblastoma
Brief Title: Efficiency of Vaccination with Lysate-loaded Dendritic Cells in Patients with Newly Diagnosed Glioblastoma
Acronym: GlioVax
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GlioVax
Record Dates: First submitted 2017-10-26; First posted 2018-01-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma
Keywords: glioblastoma,; immunotherapy; dendritic cells; vaccination
MeSH Terms: conditions — Glioblastoma | interventions — Standard of Care; Temozolomide

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, open-label, randomized phase 2 study with two parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental intervention (Experimental): Fluorescence-guided surgery (day 0) Leukapheresis (wk4) Fractionated radiotherapy (60 Gy: 2 Gy/d, 5/7 d, 6 wks; wk5 10) and concomitant TMZ chemotherapy (75 mg/m2/d; 6 wks; wk5-10) vaccination with autologous, tumor lysate-loaded, mature dendritic cells (DC) (7x, 2 - 10 x 106 DC each, intradermal injection, weekly wk11-14, wk17, 21, 25)Adjuvant TMZ chemotherapy (150-200 mg/m2/d, 6x, days 1 5 of 28 d cycle: wk15, 19, 23, 27, 31, 35)
  Interventions: Biological: Autologous, tumor lysate-loaded, mature dendritic cells (DC)
- Control intervention (Other): Standard therapy:
  Fluorescence-guided surgery (day 0) Fractionated radiotherapy (60 Gy: 2 Gy/d, 5/7 d, 6 wks; wk5 10) and concomitant TMZ chemotherapy (75 mg/m2/d; 6 wks; wk5-10) Adjuvant TMZ chemotherapy (150-200 mg/m2/d, 6x, days 1 5 of 28 d cycle: wk15, 19, 23, 27, 31, 35)
  Interventions: Drug: standard therapy

INTERVENTIONS:
Biological: Autologous, tumor lysate-loaded, mature dendritic cells (DC) — Advanced therapy medicinal product (ATMP) produced at the University Hospital Düsseldorf according to Good Manufacturing Practice (GMP) with production permission according §13 AMG (German Drug Law) of the local authorities (Bezirks¬regierung Düsseldorf)
  Other Names: dendritic cell vaccination
  Arms: Experimental intervention
Drug: standard therapy — temozolomide, fractionated radiochemotherapy
  Other Names: temozolomide, fractionated radiochemotherapy
  Arms: Control intervention

SUMMARY:
The primary objective of the study is to determine whether overall survival of newly diagnosed glioblastoma patients treated with lysate-loaded, mature dendritic cell vaccines as add-on to the standard of care consisting of resection, radiotherapy with concomitant temozolomide chemotherapy and subsequent adjuvant temozolomide chemotherapy is superior to the treatment with the standard of care alone.

DETAILED DESCRIPTION:
This is a multicenter, randomized, phase 2 study, integrating vaccination with tumorlysate-loaded mature dendritic cells into standard radio/temozolomide-chemotherapy of newly diagnosed glioblastoma patients with near-complete resection after fluorescence-guided resection. Only patients with confirmed gross-total resection and a residual tumor volume below 5 ml will be eligible for the trial. Vaccination will be performed after radio- and concomitant temozolomide chemotherapy and during the first three cycles of adjuvant TMZ.

ELIGIBILITY:
Inclusion Criteria:

Determined at pre-screening (prior to surgery; wk-3 - wk-1):

* Patients ≥ 18 years of age at surgery.
* Patients must be in a cognitive state to understand and sign the informed consent indicating that they are aware of the investigational nature and procedures of the study.
* First written informed consent for screening for eligibility, including tumor tissue collection, transfer and processing, central neuropathological evaluation of Tumor sample, central neuroradiological assessment of extent of resection, infectious disease (HIV, HBV, HCV, Treponema pallidum) testing, determination of MGMT promoter methylation status and pregnancy testing.

Determined at screening (at and post-surgery; d0 - wk3):

* Newly diagnosed, monofocal GBM, IDH wildtype (WHO grade IV), including the histological variants of gliosarcoma and giant cell glioblastoma, confirmed by central neuropathologist according to the WHO classification of central nervous System tumors 2016. Tumors may cross into, but not beyond the corpus callosum.
* Near-complete resection (≤ 5 ml residual contrast enhancing tumor volume) confirmed by central neuroradiologist on MRI scan within 72 h postoperative; awake surgery and second look surgery are possible, if medically indicated.
* Sterile tumor sample of ≥ 150 mg with tumor cell frequency ≥ 60% as determined by central neuropathologist available for vaccine production.
* Successful production of sterile, avital tumor lysate.
* Karnofsky performance status ≥ 70%.
* Adequate hepatic (serum glutamate pyruvate transferase/alanine transaminase (SGPT/ALT), serum glutamic oxaloacetate transaminase/aspartate transaminase (SGOT/AST) and alkaline phosphatase ≤ 3-times upper limit of normal (ULN); bilirubin ≤ 1.5-times ULN) and renal functions (creatinine ≤ 1.5-times ULN).
* Adequate bone marrow function (hemoglobin ≥ 10 g/dl, thrombocytes ≥ 100,000/μl, white blood cell count ≥ 3,000/μl; neutrophil count ≥ 1,500/μl).
* Prothrombin time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6x ULN unless therapeutically warranted. International normalized ratio (INR) (in absence of anticoagulation treatment) ≤ 1.5.
* Systemic corticosteroids tapered down to ≤ 2 mg of dexamethasone or equivalent per day within 7 days postoperative (use of corticosteroids during the treatment period should be avoided, however it is possible if clinically indicated, but may require interruption of dendritic cell vaccination).
* Female patients with reproductive potential and male generative patients and their female partners must agree to be true abstinent or to use a highly effective form of contraception (pearl index < 1%) during the trial.
* Patients must be in a cognitive state to understand and sign the informed consent indicating that they are aware of the investigational nature and procedures of the study.
* Written informed consent to participate in study.

Exclusion Criteria:

determined at pre-screening (prior to surgery; wk-3 - wk-1):

* Medical history of severe acute or chronic disease with poor prognosis, e.g. severe coronary heart disease, heart failure (New York Heart Association classes III/IV), severe poorly controlled diabetes, severe mental retardation or other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
* Medical history of severe autoimmune disorder or immunodeficiency or patients with organ allograft.
* Medical history of bleeding diathesis or coagulopathy.
* Prior malignancy during the last three years except non-melanoma skin cancer, in situ cervical cancer, treated superficial bladder cancer or cured, early-stage prostate cancer in a patient with prostate-specific antigen (PSA) level less than ULN.
* Previous radiotherapy to head and neck.
* Known allergy or intolerability to TMZ, dacarbazine, the contrast agent or to components of the dendritic cell vaccine.
* Current treatment of glioblastoma in another clinical trial with therapeutic intervention or current use of any other investigational agent.
* Known pregnancy or breast feeding.
* No known severe infection requiring treatment.
* Accommodation in an institution due to legal orders (§40(4) AMG).
* Evidence of current drug or alcohol abuse. determined at screening (at and post-surgery; d0 - wk3):
* Infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or Treponema pallidum or other severe infection requiring treatment.
* Accommodation in an institution due to legal orders (§40(4) AMG).
* Pregnant or breast feeding female patients. From pre-menopausal female patients with childbearing potential a negative pregnancy test must be obtained.
* Any psycho-social condition hampering compliance with the study protocol.
* MGMT promoter methylation status equivocal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Day of surgery until death of any cause assessed up to 34 months
  Overall survival as measured from the day of surgery until death from any cause assessed up to 34 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | Day of surgery until day of diagnosis of tumor progression assessed upto 34 months
  Progression-free survival as measured from the day of surgery until diagnosis of tumor progression by MRI scan according to modified Response Assessment in Neuro-Oncology (RANO) criteria assessed up to 34 months
OS rates | 6, 12 and 24 months after the day of surgery
  OS rates at 6, 12 and 24 months after the day of surgery
PFS rates | 6, 12 and 24 months after the day of surgery
  PFS rates at 6, 12 and 24 months after the day of surgery
Frequency and severity of adverse events | 34 months
  Safety based on the frequency and severity of adverse events (AE) with toxicity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events 4.03 (CTCAE 4.03)
Karnofsky Performance Status | 34 months
  Overall and neurological performance based on the Karnofsky performance status (MMSE-2)
MMSE-2 | 34 months
  Overall and neurological performance based on the Minimal Mental State Examination 2 (MMSE-2)
Quality of life of cancer patients | 34 months
  Quality of life as determined by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30 3.0
Quality of life in patients with brain cancer | 34 months
  Quality of life as determined by the European Organization for Research and Treatment of Cancer (EORTC) Brain Cancer Module QLQ-BN20
Psychological distress in oncology patients | 34 months
  Quality of life as determined by the Distress Thermometer (DT)
Psychological distress, anxiety and depression | 34months
  Quality of life as determined by the Hospital Anxiety and Depression Scale (HADS) for psycho-oncological strain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sabel, Prof. MD, Principal Investigator — Department of Neurosurgery
Locations (6):
- Germany (6):
  - Klinik für Neurologie, Knappschaftskrankenhaus Bochum, Bochum, North Rhine-Westphalia
  - Klinik für Neurochirurgie, Sana Kliniken Duisburg, Duisburg, North Rhine-Westphalia
  - Neurochirurgische Klinik, Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - St. Marien Hospital Lünen, Klinik für Neurochirurgie, Lünen, North Rhine-Westphalia
  - Klinik für Allgemeine Neurologie, Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Helios Klinikum Krefeld, Klinik für Neurochirurgie, Krefeld

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naulaerts S, Datsi A, Borras DM, Antoranz Martinez A, Messiaen J, Vanmeerbeek I, Sprooten J, Laureano RS, Govaerts J, Panovska D, Derweduwe M, Sabel MC, Rapp M, Ni W, Mackay S, Van Herck Y, Gelens L, Venken T, More S, Bechter O, Bergers G, Liston A, De Vleeschouwer S, Van Den Eynde BJ, Lambrechts D, Verfaillie M, Bosisio F, Tejpar S, Borst J, Sorg RV, De Smet F, Garg AD. Multiomics and spatial mapping characterizes human CD8+ T cell states in cancer. Sci Transl Med. 2023 Apr 12;15(691):eadd1016. doi: 10.1126/scitranslmed.add1016. Epub 2023 Apr 12. PMID 37043555
- [Derived] Rapp M, Grauer OM, Kamp M, Sevens N, Zotz N, Sabel M, Sorg RV. A randomized controlled phase II trial of vaccination with lysate-loaded, mature dendritic cells integrated into standard radiochemotherapy of newly diagnosed glioblastoma (GlioVax): study protocol for a randomized controlled trial. Trials. 2018 May 25;19(1):293. doi: 10.1186/s13063-018-2659-7. PMID 29801515